CLINICAL TRIAL: NCT00157170
Title: The Effects of a Supervised Exercise Program on Self Efficacy, Quality of Life Status, Cardiovascular Fitness and Hospital Readmission Rates of People Living With HIV/AIDS.
Brief Title: The Effects of a Supervised Exercise Program on Self Efficacy of People Living With HIV/AIDS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 92/02
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-10-21 (Estimated); Status verified 2005-05

CONDITIONS: HIV Infections
Keywords: exercise; self efficacy; quality of life; HIV
MeSH Terms: conditions — HIV Infections; Motor Activity

INTERVENTIONS:
Behavioral: supervised exercise

SUMMARY:
To evaluate the impact of a supervised exercise program (SEP) on self-efficacy,quality of life status and cardiovascular fitness among people with HIV in a 24 week randomised controlled trial.We hypothesised that a combined aerobic and resisted exercise (intervention) would improve these parameters compared to an individual walking program with monthly group forum (control).

DETAILED DESCRIPTION:
With combination antiretroviral therapy, HIV has become a chronic, manageable medical condition. Medication adherence is now a critical determinant of patient outcomes. Quality of life (QOL) rather than just survival has also become an important consideration in HIV management strategies. The role of non-pharmacological interventions such as exercise to enhance self efficacy (which correlates with adherence) and QOL among people with HIV requires formal investigation.

We evaluated the impact of a supervised exercise program (SEP) on self-efficacy among people with HIV in a 24 week, randomised controlled trial of participation in a SEP with combined aerobic and resisted exercise (intervention) versus an individual walking program with monthly group forum (control). QOL and cardiovascular fitness were also evaluated as secondary endpoints. Twenty subjects were enrolled in each arm, and assessments were performed at baseline, 2 month and 6 months, including a Generic Self Efficacy Scale, 1 minute heart rate response post 3 minute step test, and a validated HIV-specific QOL survey.

Self efficacy and cardiovascular fitness improved in the intervention but not the control subjects over the study period (p<0.0001 for both). QOL also improved (8 out of 10 dimensions) in the intervention group but not in controls (0 out of 10 dimensions).

These data support the use of SEP as an important therapeutic intervention for people with HIV, with significant benefits to self efficacy, cardiovascular fitness and QOL over six months. Importantly, these benefits were not achieved through unsupervised exercise over the same period.

ELIGIBILITY:
Inclusion Criteria:

HIV, aged at least 18 years

Exclusion Criteria:

* any contraindications to exercise testing and training , severe cognitive impairment
* inability to follow instructions,
* regular exercise ( participating in 2 or more structured exercise sessions weekly for more than or equal to 6 months prior to enrolment).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-09; Study Completion 2005-05

PRIMARY OUTCOMES:
All outcomes measured at baseline, 2 and 6 months.Self-efficacy measured by the General Self-Efficacy(GSE) Scale.

SECONDARY OUTCOMES:
Quality of life measured by MOS-HIV Scale. Cardiovascular fitness measured by the Kasch Pulse Recovery Test.

CONTACTS AND LOCATIONS:
Overall Officials: Soula Fillipas, BPhysio MPH, Principal Investigator — Bayside Health
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia